CLINICAL TRIAL: NCT06667297
Title: Correlation Between Acute Gastrointestinal Injury and Venous Return in Critical Ill Patients
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 216-3
Record Dates: First submitted 2024-01-17; First posted 2024-10-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Gastrointestinal Injury; Critical Illness
Keywords: Acute gastrointestinal injury; Venous Excess Ultrasound Score
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, altered intestinal blood flow in critically ill patients has been a hot research topic in recent years. In 2022, studies on acute mesenteric ischemia were published in top journals in critical care medicine [Crit Care, 2022. 26(1): p.92. and Intensive Care Med, 2022. 26(2): p.92.].

However, because the gastrointestinal tract is in the abdominal cavity and doctors lack methods to directly monitor the visceral perfusion. Therefore, there is little research on the relationship between gastrointestinal perfusion and acute gastrointestinal injury in critical ill patients. Currently, the diagnosis of acute gastrointestinal injury is mostly performed using subjective indicators and adverse outcomes that have already occurred, which results in the treatment of acute gastrointestinal injury often lagging behind.

The use of color Doppler ultrasonography to assess blood flow in intestinal vessels in healthy and outpatient patients has been in use since the 1980s. Our team showed that the resistance index of the superior mesenteric artery(SMA) in postoperative cardiac surgery patients correlated with lactate values and lactate clearance [Front Med (Lausanne), 2021.8: p.762376.], suggesting that gastrointestinal perfusion as reflected by SMA blood flow is important for systemic resuscitation, and that Doppler indices of SMA have the potential value of reflecting intestinal hypo-perfusion.

Intestinal venous blood enters the portal vein and then the liver before returning to the right heart via the inferior vena cava. Right ventricular dysfunction or abdominal hypertension could cause obstruction of portal venous return, which might lead to edema and dysfunction of the intestine.

Therefore, monitoring the venous return status is crucial for intestinal perfusion.

In 2012, the Venous Excess Ultrasound Score(VExUS) for evaluating venous return has been reported and it has been shown to correlate with acute kidney injury (AKI) [Intensive Care Med, 2012. 38(3): p.384-94]. However, there is currently no research on the correlation between acute gastrointestinal injury and venous return, and this study is innovative and exploratory.

DETAILED DESCRIPTION:
Research Methods

1. The Venous Excess Ultrasound Score(VExUS):

   Blood flow parameters were measured by two ICU physicians and the mean values were recorded. Both ICU physicians had more than 4 years of experience in critical care ultrasound; they were certified by the Chinese Critical Care Ultrasound Study Group. Monitoring the status of venous return in the portal vein, hepatic vein, intra-renal vein.

   The status of venous returnwere evaluated in categorical variables as normal, mildly abnormal, or severely abnormal, as previously reported. Patients were then classified according to the assessment in Grades 0-3: Grade 0, no congestion; Grade 1, mild congestion; Grade 2, moderate congestion; and Grade 3, severe congestion.To minimize errors, it is important to take the average of three measurements in a magnified state.
2. Ultrasound score of transabdominal bowel function (AGUIS score) At the time of the ultrasound examination, the operator categorized the situation as "good quality", "poor quality" or "not assessable". The abdomen is then divided into four quadrants, each measuring one point, and the operator examines and scores the diameter of the bowel, changes in bowel folds (e.g., shortening, decreasing), thickness of the bowel wall, layering of the bowel wall, peristalsis, and movement of bowel contents. A total of four scores are obtained, and the average of the four measurements is the (AGIUS) score.
3. Gastrointestinal Dysfunction Score (GIDS): 0 score (No risk): No symptoms OR one of the following with oral intake: Absent bowel sounds; Vomiting; GRV >200 mL; GI paralysis/dynamic ileus; Abdominal distension; Diarrhea (not severe); GI bleeding without transfusion; IAP >20 mmHg. 1 score(Increased risk): Two of the following: No oral intake; Absent bowel sounds; Vomiting; GRV >200 mL; GI paralysis/dynamic ileus; Abdominal distension; Diarrhea (not severe); GI bleeding without transfusion; IAP >20 mmHg. 2 score(gastrointestinal dysfunction): Three or more symptoms of score 1 OR up to two of the following: Severe diarrhea; GI bleeding with transfusion; IAP >20 mmHg. 3 score(gastrointestinal failure): Three or more of the following: Prokinetic use; GI paralysis/dynamic ileus; Abdominal distension; Severe diarrhea; GI bleeding with transfusion; IAP >20 mmHg. 4 score(Life threatening): One of the following: GI bleeding leading to hemorrhagic shock; Mesenteric ischemia; Abdominal compartment syndrome
4. Serologic indices of intestinal mucosal epithelial injury Plasma citrulline, plasma intestinal fatty acid binding protein, and D-lactic acid were measured by ELISA. (R&D Systems, Minneapolis, USA). Peripheral blood specimens were obtained and centrifuged, and the resulting plasma was frozen at -20°C and sent to the laboratory for analysis within 1 week.

Study Route:

On the day of enrollment, patients' hemodynamic parameters, measurement of VExUS, AGUIS score, GIDS score and serum specimen were recorded. Measurement of the above parameters was repeated at Day 1(ICU admission)，Day 2(between 24 and 48 h)，Day 3(between 48 and 72 h)，and Departure Day(ICU discharge).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sepsis with an expected ICU stay of more than 3 days.
2. ≥18 years of age and <80 years of age.

Exclusion Criteria:

1. Severe mesenteric or abdominal artery stenosis;
2. Fixed body (such as recent spinal surgery or intracranial hypertension);
3. Patients with contraindications for IAP measurement (such as patients who have recently undergone bladder surgery, been injured, or become pregnant）
4. Having undergone abdominal surgery or chest lowering involving the intestines patients undergoing aortic surgery;
5. Poor quality of abdominal ultrasound images;
6. Hydrothorax or ascites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU admitted patients in comprehensive hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The Venous Excess Ultrasound Score | Day 1(ICU admission)，Day 2(between 24 and 48 h)，Day 3(between 48 and 72 h)，Departure Day(ICU discharge)
  The study primary endpoint was the VExUS score. It was calculated four times during the ICU stay: within 24 h of ICU admission, after day 1 (between 24 and 48 h), after day 2 (between 48 and 72 h), and at ICU discharge. The patients were classified as being congestive (VExUS≥2) or not being congestive (VExUS < 2). A VExUS grade 2 was defined as moderate congestion, and a VExUS grade 3 was defined as severe congestion.

SECONDARY OUTCOMES:
Serologic indices of intestinal mucosal epithelial injury Plasma citrulline, plasma intestinal fatty acid binding protein, and D-lactic acid | Day 1(ICU admission)，Day 2(between 24 and 48 h)，Day 3(between 48 and 72 h)，Departure Day(ICU discharge)
  Those indices were measured by ELISA. (R&D Systems, Minneapolis, USA). Peripheral blood specimens were obtained and centrifuged, and the resulting plasma was frozen at -20°C and sent to the laboratory for analysis within 1 week
Acute gastrointestinal injury | Day 1(ICU admission)，Day 2(between 24 and 48 h)，Day 3(between 48 and 72 h)，Departure Day(ICU discharge)
  The severity of acute gastrointestinal injury is classified based on the American Association for the Surgery of Trauma (AAST) grading system. The system assigns grades from I to V, with I being the least severe and V being the most severe. Grade I injuries involve minimal damage to the mucosa and submucosa of the gastrointestinal tract. Grade II injuries involve damage to the muscularis propria layer. Grade III injuries involve damage to all layers of the gastrointestinal wall, but there is no perforation or major organ dysfunction. Grade IV injuries involve perforation or major organ dysfunction. Grade V injuries are associated with necrotic bowel or mesenteric ischemia.
GIDS | Day 1(ICU admission)，Day 2(between 24 and 48 h)，Day 3(between 48 and 72 h)，Departure Day(ICU discharge)
  a new Gastrointestinal Dysfunction Score (GIDS) for critically ill patients based on the rationale of the previously developed AGI grading system, which is similarly divided into five grades(from 0 to 4). 0=No risk ;1=Increased risk ;2=gastrointestinal dysfunction; 3= gastrointestinal failure; 4=Life threatening.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine of pekin union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No